CLINICAL TRIAL: NCT05999448
Title: Optimizing a Personalized Health Approach for Virtually Treating High-risk Caregivers During COVID-19 and Beyond
Brief Title: Promoting the Well Being of Caregivers Via Telehealth
Acronym: WellCAST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Purdue University (Other)
Collaborators: University of Virginia (Other); University of Oregon (Other); University of Canterbury (Other); University of Missouri-Columbia (Other); Indiana University (Other); Georgia State University (Other)
Responsible Party: Principal Investigator, KelleherLab, Associate Professor, Purdue University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: R01HD105502 (NIH)
Record Dates: First submitted 2023-07-17; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Caregivers; Parents
MeSH Terms: interventions — Acceptance and Commitment Therapy; Population Groups

STUDY DESIGN:
Intervention Model Description: For Waves I-II, caregivers are randomly assigned to either (1) route to a treatment using their personalized health data ("Algorithm 1") OR route to treatment randomly ("No Algorithm"); for Waves III and IV, caregivers are randomly assigned to Algorithm 1 or an optimized Algorithm 2 (Wave III) or Algorithm 2 or an optimized and final Algorithm 3 (Wave IV).
  Across Waves I-IV, caregivers are randomly assigned to receive peer coaching ("Peer Coaching") or to receive check-ins by a staff member unfamiliar with the peer coaching protocol ("No Peer Coaching").
  Across Waves I-III, a subset of caregivers are assigned to a waitlist control that does not include any treatment or peer coaching.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Care providers will be masked to the status of peer coaching and algorithm assignment. Peer coaches will be masked to the status of algorithm assignment. Data managers and statisticians evaluating study outcomes will be provided de-identified data and will not be involved in treatment-related study operations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- No Algorithm + Participation Enhancement Intervention (Experimental): Participants are randomly assigned to support program without use of a personalized health algorithm AND receive the participation enhancement intervention.
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT); Behavioral: Culturally Informed Cognitive Behavioral Therapy (CICBT), Individual; Behavioral: Culturally Informed Cognitive Behavioral Therapy (CICBT), Group; Behavioral: Dialectical Behavioral Therapy (DBT); Behavioral: Durand Sleep Intervention; Behavioral: RUBI Intervention; Behavioral: Naturalistic Communication Intervention (NCI); Behavioral: Self-Guided Resources; Behavioral: Participation Enhancement Intervention (PEI)
- No Algorithm + No Participation Enhancement Intervention (Experimental): Participants are randomly assigned to support program without use of a personalized health algorithm AND do not receive the participation enhancement intervention.
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT); Behavioral: Culturally Informed Cognitive Behavioral Therapy (CICBT), Individual; Behavioral: Culturally Informed Cognitive Behavioral Therapy (CICBT), Group; Behavioral: Dialectical Behavioral Therapy (DBT); Behavioral: Durand Sleep Intervention; Behavioral: RUBI Intervention; Behavioral: Naturalistic Communication Intervention (NCI); Behavioral: Self-Guided Resources
- Algorithm 1 + Participation Enhancement Intervention (Experimental): Participants are assigned to support programs using Algorithm 1 AND receive the participation enhancement intervention.
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT); Behavioral: Culturally Informed Cognitive Behavioral Therapy (CICBT), Individual; Behavioral: Culturally Informed Cognitive Behavioral Therapy (CICBT), Group; Behavioral: Dialectical Behavioral Therapy (DBT); Behavioral: Durand Sleep Intervention; Behavioral: RUBI Intervention; Behavioral: Naturalistic Communication Intervention (NCI); Behavioral: Self-Guided Resources; Behavioral: Participation Enhancement Intervention (PEI)
- Algorithm 1 + No Participation Enhancement Intervention (Experimental): Participants are assigned to support programs using Algorithm 1 AND do not receive the participation enhancement intervention.
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT); Behavioral: Culturally Informed Cognitive Behavioral Therapy (CICBT), Individual; Behavioral: Culturally Informed Cognitive Behavioral Therapy (CICBT), Group; Behavioral: Dialectical Behavioral Therapy (DBT); Behavioral: Durand Sleep Intervention; Behavioral: RUBI Intervention; Behavioral: Naturalistic Communication Intervention (NCI); Behavioral: Self-Guided Resources
- Algorithm 2 + Participation Enhancement Intervention (Experimental): Participants are assigned to support programs using Algorithm 2 AND receive the participation enhancement intervention.
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT); Behavioral: Culturally Informed Cognitive Behavioral Therapy (CICBT), Individual; Behavioral: Culturally Informed Cognitive Behavioral Therapy (CICBT), Group; Behavioral: Dialectical Behavioral Therapy (DBT); Behavioral: Durand Sleep Intervention; Behavioral: RUBI Intervention; Behavioral: Naturalistic Communication Intervention (NCI); Behavioral: Self-Guided Resources; Behavioral: Participation Enhancement Intervention (PEI)
- Algorithm 2 + No Participation Enhancement Intervention (Experimental): Participants are assigned to support programs using Algorithm 2 AND do not receive the participation enhancement intervention.
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT); Behavioral: Culturally Informed Cognitive Behavioral Therapy (CICBT), Individual; Behavioral: Culturally Informed Cognitive Behavioral Therapy (CICBT), Group; Behavioral: Dialectical Behavioral Therapy (DBT); Behavioral: Durand Sleep Intervention; Behavioral: RUBI Intervention; Behavioral: Naturalistic Communication Intervention (NCI); Behavioral: Self-Guided Resources
- Algorithm 3 + Participation Enhancement Intervention (Experimental): Participants are assigned to support programs using Algorithm 3 AND receive the participation enhancement intervention.
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT); Behavioral: Culturally Informed Cognitive Behavioral Therapy (CICBT), Individual; Behavioral: Culturally Informed Cognitive Behavioral Therapy (CICBT), Group; Behavioral: Dialectical Behavioral Therapy (DBT); Behavioral: Durand Sleep Intervention; Behavioral: RUBI Intervention; Behavioral: Naturalistic Communication Intervention (NCI); Behavioral: Self-Guided Resources; Behavioral: Participation Enhancement Intervention (PEI)
- Algorithm 3 + No Participation Enhancement Intervention (Experimental): Participants are assigned to support programs using Algorithm 3 AND do not receive the participation enhancement intervention.
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT); Behavioral: Culturally Informed Cognitive Behavioral Therapy (CICBT), Individual; Behavioral: Culturally Informed Cognitive Behavioral Therapy (CICBT), Group; Behavioral: Dialectical Behavioral Therapy (DBT); Behavioral: Durand Sleep Intervention; Behavioral: RUBI Intervention; Behavioral: Naturalistic Communication Intervention (NCI); Behavioral: Self-Guided Resources
- Waitlist Control (No Intervention): Participants are enrolled in the waitlist control condition, which includes identical data collection procedures to participants enrolled in support programs. Waitlist controls are offered the opportunity to enroll in future cycles.

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy (ACT) — ACT will be deployed weekly for 12 weeks on an individual basis via secure Zoom. Treatments will be deployed by supervised graduate student clinicians under the supervision of a licensed psychologist.
  Arms: Algorithm 1 + No Participation Enhancement Intervention; Algorithm 1 + Participation Enhancement Intervention; Algorithm 2 + No Participation Enhancement Intervention; Algorithm 2 + Participation Enhancement Intervention; Algorithm 3 + No Participation Enhancement Intervention; Algorithm 3 + Participation Enhancement Intervention; No Algorithm + No Participation Enhancement Intervention; No Algorithm + Participation Enhancement Intervention
Behavioral: Culturally Informed Cognitive Behavioral Therapy (CICBT), Individual — CICBT-Individual will be deployed weekly for 12 weeks on an individual basis via secure Zoom. Treatments will be deployed by supervised graduate student clinicians under the supervision of a licensed psychologist.
  Other Names: Trauma Focused Cognitive Behavioral Therapy
  Arms: Algorithm 1 + No Participation Enhancement Intervention; Algorithm 1 + Participation Enhancement Intervention; Algorithm 2 + No Participation Enhancement Intervention; Algorithm 2 + Participation Enhancement Intervention; Algorithm 3 + No Participation Enhancement Intervention; Algorithm 3 + Participation Enhancement Intervention; No Algorithm + No Participation Enhancement Intervention; No Algorithm + Participation Enhancement Intervention
Behavioral: Culturally Informed Cognitive Behavioral Therapy (CICBT), Group — CICBT-Group will be deployed weekly for 12 weeks in small groups via secure Zoom. Treatments will be deployed by supervised graduate student clinicians under the supervision of a licensed psychologist.
  Other Names: Trauma Focused Cognitive Behavioral Therapy
  Arms: Algorithm 1 + No Participation Enhancement Intervention; Algorithm 1 + Participation Enhancement Intervention; Algorithm 2 + No Participation Enhancement Intervention; Algorithm 2 + Participation Enhancement Intervention; Algorithm 3 + No Participation Enhancement Intervention; Algorithm 3 + Participation Enhancement Intervention; No Algorithm + No Participation Enhancement Intervention; No Algorithm + Participation Enhancement Intervention
Behavioral: Dialectical Behavioral Therapy (DBT) — DBT will be deployed weekly for 12 weeks in small groups via secure Zoom. Treatments will be deployed by supervised graduate student clinicians under the supervision of a licensed psychologist.
  Arms: Algorithm 1 + No Participation Enhancement Intervention; Algorithm 1 + Participation Enhancement Intervention; Algorithm 2 + No Participation Enhancement Intervention; Algorithm 2 + Participation Enhancement Intervention; Algorithm 3 + No Participation Enhancement Intervention; Algorithm 3 + Participation Enhancement Intervention; No Algorithm + No Participation Enhancement Intervention; No Algorithm + Participation Enhancement Intervention
Behavioral: Durand Sleep Intervention — Durand Sleep Intervention will be deployed weekly for 12 weeks, alternating between individual and group formats, via secure Zoom. Treatments will be deployed by supervised graduate student clinicians under the supervision of a licensed psychologist or behavioral analyst.
  Arms: Algorithm 1 + No Participation Enhancement Intervention; Algorithm 1 + Participation Enhancement Intervention; Algorithm 2 + No Participation Enhancement Intervention; Algorithm 2 + Participation Enhancement Intervention; Algorithm 3 + No Participation Enhancement Intervention; Algorithm 3 + Participation Enhancement Intervention; No Algorithm + No Participation Enhancement Intervention; No Algorithm + Participation Enhancement Intervention
Behavioral: RUBI Intervention — RUBI will be deployed weekly for 12 weeks in small groups via secure Zoom. Treatments will be deployed by supervised graduate student clinicians under the supervision of a licensed behavioral analyst.
  Arms: Algorithm 1 + No Participation Enhancement Intervention; Algorithm 1 + Participation Enhancement Intervention; Algorithm 2 + No Participation Enhancement Intervention; Algorithm 2 + Participation Enhancement Intervention; Algorithm 3 + No Participation Enhancement Intervention; Algorithm 3 + Participation Enhancement Intervention; No Algorithm + No Participation Enhancement Intervention; No Algorithm + Participation Enhancement Intervention
Behavioral: Naturalistic Communication Intervention (NCI) — NCI will be deployed weekly for 12 weeks on an individual basis via secure Zoom. Treatments will be deployed by supervised graduate student clinicians under the supervision of a licensed behavioral analyst.
  Arms: Algorithm 1 + No Participation Enhancement Intervention; Algorithm 1 + Participation Enhancement Intervention; Algorithm 2 + No Participation Enhancement Intervention; Algorithm 2 + Participation Enhancement Intervention; Algorithm 3 + No Participation Enhancement Intervention; Algorithm 3 + Participation Enhancement Intervention; No Algorithm + No Participation Enhancement Intervention; No Algorithm + Participation Enhancement Intervention
Behavioral: Self-Guided Resources — Participants will be provided a self-guided resource notebook that includes 12 weeks of content that parallels the topics examined in other support programs (child behavior management, child sleep, child communication, caregiver mental health, caregiver health behaviors, community connection)
  Arms: Algorithm 1 + No Participation Enhancement Intervention; Algorithm 1 + Participation Enhancement Intervention; Algorithm 2 + No Participation Enhancement Intervention; Algorithm 2 + Participation Enhancement Intervention; Algorithm 3 + No Participation Enhancement Intervention; Algorithm 3 + Participation Enhancement Intervention; No Algorithm + No Participation Enhancement Intervention; No Algorithm + Participation Enhancement Intervention
Behavioral: Participation Enhancement Intervention (PEI) — A standardized PEI intervention will be conducted by trained peer coaches who are also rare disorder caregivers. Each peer coach will work with their clients to complete a "Change Plan Worksheet" and will complete two booster sessions at midpoint and end of treatment. Coaches will also meet with their clients after follow-up data are complete to support connection back to community resources and patient-specific rare disorder communities.
  Arms: Algorithm 1 + Participation Enhancement Intervention; Algorithm 2 + Participation Enhancement Intervention; Algorithm 3 + Participation Enhancement Intervention; No Algorithm + Participation Enhancement Intervention

SUMMARY:
The goal of this clinical trial is to learn which types of telehealth-based treatments best fit the needs of caregivers of people with rare neurogenetic conditions. The main questions it plans to answer are:

* Which telehealth support programs best meet the needs of rare disorder caregivers?
* How can individuals be matched to support programs that are right for them? What aspects of an individual (e.g., demographics, mental health symptoms, family characteristics, lifestyle) predict whether treatment will be a good fit?
* Does peer-to-peer coaching help improve patients' experiences during telehealth treatment?

Participants will be asked to complete a 12-week treatment program, which may include self-guided resources, individual therapies, group therapies, and/or peer-to-peer coaching.

Before, during, and after treatment, participants will complete questionnaires to help researchers understand their experiences, symptoms, and impressions of their support program. Questionnaires will include both standard forms (administered up to 5 times throughout the study) and brief "snapshot surveys" that participants complete on their smartphones up to 3 times per day.

Some participants will be assigned to a waitlist control, which means that they will provide data while they are not yet completing a support program. These participants will be assigned to a support program in the next treatment phase.

DETAILED DESCRIPTION:
Project WellCAST (Supporting Wellbeing of Caregivers via Telehealth) is a multi-phase research study that aims to develop a scalable, personalized health approach for supporting caregivers of people with rare disorders. Two previous studies by this research team have piloted individual interventions in subsets of rare disorder caregiving communities to establish initial feasibility and acceptability. Now in its third phase, Project WellCAST 3.0 aims to generate a scalable, innovative model for personalizing digital treatments to caregiver needs. This project has two specific aims:

AIM 1: Develop and optimize a personalized health algorithm to match neurogenetic syndrome (NGC) caregivers to digital health treatments using a combination of standard clinical tools and smartphone-based EMA data.

Extant clinical and EMA data on NGC caregiver response to COVID-19 was used to develop an initial routing algorithm to match families to treatment type and intensity. This aim will compare the effectiveness of algorithm-assigned treatment to "treatment as usual," optimizing the algorithm across four waves of intervention. Interventions will be brief, evidence-based, digital health treatments administered by highly supervised clinical trainees, a cost-efficient model for directly targeting the secondary health effects of COVID-19.

AIM 2: Test the efficacy of peer-to-peer coaching, deployed by trained NGC caregivers using an evidence-based motivational interviewing protocol, in enhancing treatment uptake and clinical outcomes.

Peer coaches who are also NGC caregivers will be trained to deploy evidence-based Participation Enhancement Interventions designed to support treatment engagement and reduce potential barriers. This aim will evaluate the feasibility and effectiveness of this approach in reducing secondary health effects of COVID-19 by comparing outcomes across participants who were randomized to complete treatment with and without peer coaches. Peer coaches will also provide valuable stakeholder input for designing and optimizing the digital treatment network.

DETAILED HUMAN SUBJECTS PROCEDURE:

ENROLLMENT AND CONSENT 1. At the entry of the study, caregivers will be assessed by the study team to determine eligibility. The caregivers will then consent to baseline collection. A subset of caregivers will be enrolled at this phase as waitlist controls. Waitlist controls will complete the same data collection described below, but without any support program.

BASELINE. The baseline period of the study lasts two weeks. During this time, caregivers will complete initial study forms and "snapshot surveys," which are brief questionnaires sent three times per day via their smartphones.

ROUTING. After baseline data collection is complete, caregivers will be routed to a support program. Random number generators will be used to route caregivers to their study arm, described below.

Caregivers may opt out of broadly completing either child-focused or self-focused treatments but may not select their specific treatment modality. As an exception, any Black caregiver in the study is eligible to add the CICBT group to their assigned support program.

CONSENT 2 and INTERVENTION. Participants will provide informed consent specific to their assigned intervention then begin their 12-week support program. Programs are described below. During intervention, caregivers will be asked to complete study forms to assess how their characteristics and experiences have changed interventions; forms will be collected at start of treatment, midpoint, and endpoint. Caregivers will also complete "snapshot surveys" (3x/day) during this time.

FOLLOW UP. Two weeks after completing treatment, caregivers will complete follow-up forms and a 2-week period of "snapshot surveys."

ADDITIONAL PROCEDURES:

This study will occur across four phases. Phases I and II will enroll up to 500 participants (to yield 400 participants total) who will be randomly assigned to Algorithm (Algorithm 1 versus No Algorithm) and Peer Coaching (Peer Coaching versus No Peer Coaching).

After Phase II, investigators will convene a "think tank" that will evaluate primary and secondary endpoints across arms, with the goal of determining how to optimize the algorithm. Data analyses will be performed by staff who are not involved in clinical operations. Peer coaches (who are rare disorder caregivers), clinicians, biostatisticians, and scientists will collaboratively participate in this think tank, with the goal to optimize the algorithm prior to Phase III.

Phase III will enroll up to 250 participants (to yield 200) who will receive the optimized Algorithm 2 and be randomly assigned to Peer Coaching conditions. After Phase III, a second think tank will be convened to optimize Algorithm 3.

Phase IV will enroll up to 250 participants (to yield 200) who will receive the optimized Algorithm 3 and will be randomly assigned to Peer Coaching conditions.

Final analyses will compare Algorithm 3 to Algorithm 2, Algorithm 1, and Waitlist Controls.

RIGOR AND REPRODUCIBILITY.

Algorithms will be uploaded to a secure, locked site prior to each round of study assignment. Analyses will be preregistered, and all code will be available for replication efforts. Masking procedures are described elsewhere in this document.

ELIGIBILITY:
Inclusion Criteria:

* Caregiver and legal guardian of child age 2-35 with neurogenetic condition
* Child's syndrome must (1) have an established genetic cause, (2) affect the brain, resulting in moderate to severe intellectual disability in the majority of patients
* Reside in US
* Fluent in English (spoken and written)
* Seeking support for caregiver mental health/well-being and/or caregiving needs

Exclusion Criteria:

* Serious mental illness or active addiction that would be inadequately addressed through dosage of treatments
* Actively in treatment that would be redundant with those offered in the protocol
* Child's syndrome is not commonly associated with (1) life expectancy less than 35 years or (2) deterioration of previously gained skills.

Additional treatment-specific inclusion criteria are embedded in the experimental algorithm that will be adjusted through Aim 1.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2023-06-28 (Actual); Primary Completion 2025-09-08 (Estimated); Study Completion 2025-12-29 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline on DASS-21 Total-Score at End-of-Treatment Survey | Baseline and End-of-Treatment (Treatment Week 12)
  The patient-reported Depression, Anxiety, and Stress Scale, 21 Total Score ranges from 0-63; higher scores indicate greater impairment. Change is measured as (Week 12-Baseline), statistically controlling for Baseline levels.
Change from Baseline on PSOC Total Score at End-of-Treatment Survey | Baseline and End-of-Treatment (Treatment Week 12)
  The patient-reported Parenting Sense of Competence Total Score includes ranges from 17-102; higher scores indicate greater parenting sense of competency. Wording was adapted from the original 1978 measure to be inclusive of caregivers who are not biological parents or mothers. Change is measured as (Week 12-Baseline), statistically controlling for Baseline symptoms.
Change from Baseline on PSI-4-SF Total Score at End-of-Treatment Survey | Baseline and End-of-Treatment (Treatment Week 12)
  The patient-reported Parenting Stress Index, 4th Edition (PSI-4-SF) Total T-Score ranges from 0-100; higher scores indicate greater stress. Change is measured as (Week 12-Baseline), statistically controlling for Baseline symptoms.
Change in Average PANAS Negative Affect between Baseline and End-of-Treatment | Baseline and End-of-Treatment (Treatment Week 12)
  The patient-reported Positive and Negative Affect Scale (10 items) Negative Affect subscale total score ranges from 10-50; higher scores indicate greater negative affect. For each evaluation period, scores will be averaged across week-long patient-reported ecological momentary assessments, which are collected 3 times per day and 7 days per week. Change will be measured as (Week 12-Baseline), statistically controlling for Baseline levels.
Change in Average Momentary Stress between Baseline and End-of-Treatment | Baseline and End-of-Treatment (Treatment Week 12)
  The patient-reported momentary stress item ranges from 0-100; higher scores indicate greater stress. For each evaluation period, scores will be averaged across week-long patient-reported ecological momentary assessments, which are collected 3 times per day and 7 days per week. Change will be measured as (Week 12-Baseline), statistically controlling for Baseline levels.
Change from Baseline on CGI-S at End-of-Treatment | Baseline and End-of-Treatment (Treatment Week 12)
  The Clinical Global Impression-Severity (CGI-S) is rated by the patient's primary clinician on a scale of 1-7, with higher scores indicating greater impairment. Change will be measured as (Week 12-Baseline), statistically controlling for Baseline levels.
Clinical Global Impression-Improvement (CGI-I) at End-of-Treatment | End-of-Treatment (single administration at Treatment Week 12)
  The Clinical Global Impression-Improvement (CGI-S) is rated by the patient's primary clinician on a scale of 1-7, with higher scores indicating greater impairment. Change will be measured as (Week 12-Baseline), statistically controlling for Baseline levels.
Peer Coach Fidelity Across Treatment Sessions | Calculated at End-of-Treatment (Treatment Week 12)
  Fidelity will be observer-rated by reliable coders to generate a fidelity ratio (0-100%), defined as the proportion of pre-defined critical session components administered to "acceptable" criterion; higher ratios indicate greater fidelity. The total fidelity score for each patient is calculated as the average of completed Baseline, Midpoint, and End-of-Treatment sessions.
Coaching Session Completion | Calculated at End-of-Treatment (Treatment Week 12)
  Completion will be reported by project staff and used to generate a completion ratio (0-100%), defined as the proportion of sessions attended; higher ratios indicate greater completion.
Treatment Session Completion | Calculated at End-of-Treatment (Treatment Week 12)
  Completion will be reported by clinicians to generate a completion ratio (0-100%), defined as the proportion of sessions attended; higher ratios indicate greater completion. Participants in the self-guided resource condition will self-report completion across 12 weeks of tasks using a log submitted at end of treatment.
Peer Coaching Satisfaction | End-of-Treatment (single administration at Treatment Week 12)
  Patient-reported peer coaching satisfaction scores are averaged across a study-specific feedback survey and range from 1-5; higher scores indicate greater satisfaction.
Treatment Satisfaction | End-of-Treatment (single administration at Treatment Week 12)
  Patient-reported treatment satisfaction scores are averaged across a study-specific feedback survey and range from 1-5; higher scores indicate greater satisfaction.
Drop Out Status | Calculated at End-of-Treatment (Treatment Week 12)
  "Drop out" is defined as discontinuation of treatment after consenting to treatment and attending at least one session, including active discontinuation and patients lost to follow-up. Variable is dummy coded where 0=patient did not drop out, 1=patient dropped out.
Homework Completion | Calculated at End-of-Treatment (Treatment Week 12)
  Completion will be reported by clinicians to generate a completion ratio (0-100%), defined as the proportion of assigned session homework completed; higher ratios indicate greater completion. Participants in the self-guided resource condition will self-report completion across 12 weeks of tasks using a log submitted at end of treatment.

SECONDARY OUTCOMES:
Change from Baseline on EES-2 Total Score at End-of-Treatment Survey | Baseline and End-of-Treatment (Treatment Week 12)
  The patient-reported Emotion Efficacy Scale-2 (Revised) generates a Total Score from 10-50; higher scores indicate greater emotion efficacy. Change is measured as (Week 12-Baseline), statistically controlling for Baseline symptoms.
Change from Baseline on DERS Total Score at End-of-Treatment Survey | Baseline and End-of-Treatment (Treatment Week 12)
  The patient-reported Difficulties in Emotion Regulation Scale (DERS) Total Score includes possible scores that range from 36-180; higher scores indicate greater difficulties in emotion regulation. Change is measured as (Week 12-Baseline), statistically controlling for Baseline symptoms.
Change from Baseline on CBCL Total Problem Behaviors at End-of-Treatment Survey | Baseline and End-of-Treatment (Treatment Week 12)
  The patient-rated Child Behavior Checklist (CBCL 1.5-5), which the patient uses to describe their child's behaviors, yields a Total Problem Behaviors T-Score that ranges from 50-100; higher scores indicate greater child challenging behavior. Change is measured as (Week 12-Baseline), statistically controlling for Baseline symptoms.
Change from Baseline on CDI-Words and Gestures at End-of-Treatment Survey | Baseline and End-of-Treatment (Treatment Week 12)
  The patient-rated Communicative Development Inventory, Words and Gestures Edition (Vocabulary Checklist: Level I), which the patient uses to describe their child's language, yields a yields a total raw score ranging from 0-89; higher scores indicate greater communicative development. Primary outcome will be "understanding" subscale total score. Change is measured as (Week 12-Baseline), statistically controlling for Baseline symptoms.
Change from Baseline on CSHQ at End-of-Treatment Survey | Baseline and End-of-Treatment (Treatment Week 12)
  The patient-rated Children's Sleep Habits Questionnaire, which the patient uses to describe their child's behaviors, yields a total raw score ranging from 33-99; higher scores indicate greater sleep challenges. Change is measured as (Week 12-Baseline), statistically controlling for Baseline symptoms.
Change from Baseline on Albany Sleep Problems scale at End-of-Treatment Survey | Baseline and End-of-Treatment (Treatment Week 12)
  The patient-rated Albany Sleep Problems scale, which the patient uses to describe their child's behaviors, yields a total raw score ranging from 0-164; higher scores indicate greater sleep challenges. Change is measured as (Week 12-Baseline), statistically controlling for Baseline symptoms.
Change from Baseline on ZBI-7 at End-of-Treatment Survey | Baseline and End-of-Treatment (Treatment Week 12)
  The patient-reported Zarit Burden Inventory Short Form (7 item version) generates a Total Score that ranges from 0-49; higher scores indicate greater burden. Change is measured as (Week 12-Baseline), statistically controlling for Baseline symptoms.
Change from Baseline on ABC-2 at End-of-Treatment Survey | Baseline and End-of-Treatment (Treatment Week 12)
  The patient-rated Aberrant Behavior Checklist - 2nd edition, which the patient uses to describe their child's behaviors, yields a total raw score that ranges from 0-174; higher scores indicate greater child challenging behavior. Change is measured as (Week 12-Baseline), statistically controlling for Baseline symptoms.
Change from Baseline on MIBI at End-of-Treatment Survey | Baseline and End-of-Treatment (Treatment Week 12)
  The patient-reported Multidimensional Inventory of Black Identity (MIBI) generates a Total Score that ranges from 0-49; higher scores indicate greater burden. Change is measured as (Week 12-Baseline), statistically controlling for Baseline symptoms.
Change from Baseline on PCL-5 at End-of-Treatment Survey | Baseline and End-of-Treatment (Treatment Week 12)
  The patient-reported PTSD Checklist for DSM-5 (PCL-5) generates a Total Score that ranges from 0-80; higher scores indicate greater burden. Change is measured as (Week 12-Baseline), statistically controlling for Baseline symptoms.

OTHER OUTCOMES:
Change in Daily Reports of Health Behaviors between Baseline and End-of-Treatment | Baseline and End-of-Treatment (Treatment Week 12)
  Patients report daily on prior day exercise and substance use; these values will be averaged to yield total scores between 0-100%; higher scores indicate greater proportion of days engaged in exercise and substance use, respectively. For each evaluation period, scores will be averaged across week-long data collection period; these items are collected one time per day, 7 days per week. Change will be measured as (Week 12-Baseline), statistically controlling for Baseline levels.
Change in Daily Reports of Caregiver Sleep between Baseline and End-of-Treatment | Baseline and End-of-Treatment (Treatment Week 12)
  Patients report daily on prior day sleep quality (0-100) and duration (0-24 hours); higher scores indicate greater sleep quality and duration, respectively. These items are collected one time per day, 7 days per week, and will be averaged to create one value per week. Change will be measured as (Week 12-Baseline), statistically controlling for Baseline levels.
Change in Momentary Self-Efficacy between Baseline and End-of-Treatment | Baseline and End-of-Treatment (Treatment Week 12)
  The patient-reported momentary competency item is a single rating from 0-100, and higher scores indicate greater perceptions that a person can handle their day. For each evaluation period, scores will be averaged across week-long patient-reported ecological momentary assessments, which are collected 3 times per day and 7 days per week. Change will be measured as (Week 12-Baseline), statistically controlling for Baseline levels.
Change in Daily Reports of Child Challenging Behaviors between Baseline and End-of-Treatment | Baseline and End-of-Treatment (Treatment Week 12)
  The patient-reported challenging behavior items monitor (1) severity (scale 0-100) and (2) frequency (0-4 on Likert scale), where higher scores indicate more challenging behaviors. These items are collected one time per day, 7 days per week, and will be averaged to create one value per week. Change will be measured as (Week 12-Baseline), statistically controlling for Baseline levels.

CONTACTS AND LOCATIONS:
Overall Officials: Bridgette Kelleher, PhD, Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared with other researchers using best-practices in open science.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Primary outcome IPD will be shared no later than 12 months after study completion.
Access Criteria: Data access may be requested for eligible studies and qualified researchers for the purpose of addressing specific scientific objectives. A mutually signed Data Use Agreement (non-negotiable contract for data use and sharing) must be in place before accessing requested information. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with only information necessary to address the research objectives under the terms of the data sharing agreement.

REFERENCES:
- [Derived] Kelleher BL. CASCADE: a community-engaged action model for generating rapid, patient-engaged decisions in clinical research. BMC Med Res Methodol. 2025 Jul 1;25(1):168. doi: 10.1186/s12874-025-02565-7. PMID 40597746
- [Derived] Kelleher B, Emerson K, Graham LN, Vozka V, Wheeler A, Fadel W, Foti D, Metzger I, Rispoli M, Machalicek W, McLay L, Lane S, Neo WS, Carter A, Brown L, Brown J, McIntyre LL, Salwitz E, Dietz G, Naughton R, Peek K, Hollins N, Woodford E. Optimizing a Personalized Health Approach for Virtually Treating High-Risk Caregivers of Children With Neurogenetic Conditions (Project WellCAST): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Jun 25;14:e64360. doi: 10.2196/64360. PMID 40560646
- [Derived] Kelleher BL. CASCADE: A Community-Engaged Action Model for Generating Rapid, Patient-Engaged Decisions in Clinical Research. Res Sq [Preprint]. 2024 Aug 27:rs.3.rs-4790564. doi: 10.21203/rs.3.rs-4790564/v1. PMID 39257986